CLINICAL TRIAL: NCT04145791
Title: Ice Application for Postoperative Pain: a Randomized Control Trial
Brief Title: Ice Application for Postoperative Pain
Acronym: Ice-POP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Kimberly Kho, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 072018-055
Record Dates: First submitted 2019-03-01; First posted 2019-10-31 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No Ice (No Intervention): Patients will receive standard postoperative pain control methods as defined by the participating institution
- Ice (Experimental): Patients will receive ice packs to the abdomen, in addition to standard postoperative pain control methods as defined by the participating institution
  Interventions: Other: Ice

INTERVENTIONS:
Other: Ice — ice packs
  Arms: Ice

SUMMARY:
The purpose of the proposed study is to investigate the effectiveness of cryotherapy as an additional form of pain control in women undergoing laparoscopic hysterectomy for benign gynecologic conditions through a randomized trial.

DETAILED DESCRIPTION:
The purpose of the proposed study is to investigate the effectiveness of cryotherapy as an additional form of pain control in women undergoing laparoscopic hysterectomy for benign gynecologic conditions through a randomized trial. The following aims will be pursued:

Primary Aim: To determine if cryotherapy patients will have lower pain scores on VAS compared to standard pain management patients.

Primary Hypothesis: Patients receiving cryotherapy will have lower VAS scores compared to patients receiving pain management.

Secondary Aim 1: To determine if cryotherapy will reduce the number of morphine milligram equivalent (MME) compared to patients with standard pain management.

Secondary Hypothesis 1: Patients receiving cryotherapy will have lower MME values compared to patients with standard pain management.

Secondary Aim 2: To determine if cryotherapy will result in earlier return to baseline activity as measured by Quality of Recovery Questionnaire (QoR).

Secondary Hypothesis 2: Patients receiving cryotherapy will return to baseline activity level sooner than those receiving standard pain management.

Secondary Aim 3: To determine if cryotherapy will result in a faster time to discharge as determined by duration between admission to postanesthesia care unit (PACU) and discharge home.

Secondary Hypothesis 3: Patient receiving cryotherapy will be have a shorter stay in PACU.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing laparoscopic hysterectomy for benign indications within 8 weeks of enrollment
* Women >18 years of age
* Non-emergent surgery
* Non-pregnant
* Women undergoing laparoscopic hysterectomy with the minimally invasive surgery team

Exclusion Criteria:

* Requires surgery for urinary incontinence
* Has acute angle glaucoma
* Has severe cardiac/respiratory disease
* Current chronic pain condition (ie chronic pelvic pain, fibromyalgia, chronic low back pain)
* Chronic use/abuse of opioid medications for greater than 1 week preceding procedure
* Chronic NSAID use
* Current treatment of opioid dependence with methadone or buprenorphine
* Non-English or Non-Spanish speaking
* Procedure converted to laparotomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Pain score of cryotherapy patients as compared to non-cryotherapy patients | pain score collected at admission to the preoperative holding unit prior to surgery
  To determine if cryotherapy patients will have lower pain scores on a visual analog scale (VAS) compared to standard pain management patients at the time of same day discharge. VAS requires that patients mark their level pain along a straight 100mm line. There are no number markings on the scale. The beginning of the line is labeled on the left as "no pain" and the end of the line on the right is labeled as "worst pain imaginable." Once marked by the patient, the distance from beginning of the line to the patient's hash mark is measured in millimeters and that value is recorded as the pain level. The minimum is 0 (no pain) and the maximum is 100 (worst pain imaginable).
Pain score of cryotherapy patients as compared to non-cryotherapy patients | pain score collected immediately after surgery
  To determine if cryotherapy patients will have lower pain scores on a visual analog scale (VAS) compared to standard pain management patients at the time of same day discharge. VAS requires that patients mark their level pain along a straight 100mm line. There are no number markings on the scale. The beginning of the line is labeled on the left as "no pain" and the end of the line on the right is labeled as "worst pain imaginable." Once marked by the patient, the distance from beginning of the line to the patient's hash mark is measured in millimeters and that value is recorded as the pain level. The minimum is 0 (no pain) and the maximum is 100 (worst pain imaginable).
Pain score of cryotherapy patients as compared to non-cryotherapy patients | pain score collected post operative day 1
  To determine if cryotherapy patients will have lower pain scores on a visual analog scale (VAS) compared to standard pain management patients at the time of same day discharge. VAS requires that patients mark their level pain along a straight 100mm line. There are no number markings on the scale. The beginning of the line is labeled on the left as "no pain" and the end of the line on the right is labeled as "worst pain imaginable." Once marked by the patient, the distance from beginning of the line to the patient's hash mark is measured in millimeters and that value is recorded as the pain level. The minimum is 0 (no pain) and the maximum is 100 (worst pain imaginable).
Pain score of cryotherapy patients as compared to non-cryotherapy patients | pain score collected at two weeks post operative.
  To determine if cryotherapy patients will have lower pain scores on a visual analog scale (VAS) compared to standard pain management patients at the time of same day discharge. VAS requires that patients mark their level pain along a straight 100mm line. There are no number markings on the scale. The beginning of the line is labeled on the left as "no pain" and the end of the line on the right is labeled as "worst pain imaginable." Once marked by the patient, the distance from beginning of the line to the patient's hash mark is measured in millimeters and that value is recorded as the pain level. The minimum is 0 (no pain) and the maximum is 100 (worst pain imaginable).

SECONDARY OUTCOMES:
Narcotic usage | postoperative day one
  Amount of narcotic pain medicines used as measured in morphine milligram equivalent (MME).
Quality of Recovery (QoR) | through study completion to take place at preoperative visit, and post operative day #14.
  Return to baseline activity as measured by QoR questionnaire. The questionnaire consists of 15 items, 10 in Part A and 5 in Part B. Part A assesses patients daily functioning and utilizes a Likert scale 0 to 10, where 0 = none of the time [poor] and 10 = all of the time [excellent]. Park B asses symptomatology and utilizes a Likert scale (0 to 10, where 10 = none of the time [excellent] and 0 = all of the time [poor].
Time to discharge | day of surgery, up to 1440 minutes
  Duration of time in minutes between admission to postanesthesia care unit (PACU) and discharge home as recorded in the electronic health record.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kho, MD, Principal Investigator — University of Texas as Southwestern Medical Center
Locations (2):
- United States (2):
  - Parkland Health and Hospital System, Dallas, Texas
  - Clements University Hospital, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shields JK, Kenyon L, Porter A, Chen J, Chao L, Chang S, Kho KA. Ice-POP: Ice Packs for Postoperative Pain: A Randomized Controlled Trial. J Minim Invasive Gynecol. 2023 Jun;30(6):455-461. doi: 10.1016/j.jmig.2023.01.015. Epub 2023 Feb 4. PMID 36740018